CLINICAL TRIAL: NCT06394713
Title: A Phase 1b/2 Trial to Evaluate the Efficacy and Safety of QLF31907 (PD-L1/4-1BB Bi-specific Antibody) Combination Therapy in Patients With Advanced Malignant Tumors
Brief Title: A Study to Evaluate the Efficacy and Safety of QLF31907 Combination Therapy in Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLF31907-202
Record Dates: First submitted 2024-04-22; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — Irinotecan; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLF31907 in combination with Irinotecan (Experimental)
  Interventions: Drug: QLF31907; Drug: Irinotecan
- QLF31907 in combination with Docetaxel (Experimental)
  Interventions: Drug: QLF31907; Drug: Docetaxel

INTERVENTIONS:
Drug: QLF31907 — intravenous administration, once every 3 weeks
Drug: Irinotecan — intravenous administration, 125 mg/m2, d1 and d8, every 3 weeks
  Arms: QLF31907 in combination with Irinotecan
Drug: Docetaxel — intravenous administration, 75mg/m2, d1, every 3 weeks
  Arms: QLF31907 in combination with Docetaxel

SUMMARY:
This study is designed to evaluate the safety and efficacy of QLF31907 combination therapy in advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. subjects voluntarily participated and signed a written informed consent form;
2. age ≥18 years, male or female;
3. ECOG PS 0-1;
4. histopathologically diagnosed advanced malignant tumors;
5. at least 1 measurable lesion according to RECIST v1.1 criteria or Lugano (2014) criteria;
6. adequate organ function;

Exclusion Criteria:

1. previous treatment with 4-1BB agonist or 4-1BB recombinant fusion protein;
2. received anti-tumor therapy within 4 weeks prior to the first study treatment;
3. history of autoimmune disease;
4. history of other active malignancies within 3 years prior to the first treatment;
5. history of serous cardiovascular events;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
phase Ib: Dose-limiting toxicity(DLT) | 28 days
  The DLT of QLF31907 combination therapy will be determined
phase2: objective response rate(ORR) | up to 2 years
  the ORR of QLF31907 combinaton therapy will be determined

SECONDARY OUTCOMES:
adverse events (AEs) of QLF31907 combination therapy | up to 2 years
  to evaluate the severity, incidence and causality of adverse events (AEs)
area under the concentration-time curve (AUC) of QLF31907 | up to 2 years
  the area under the concentration-time curve (AUC) of QLF31907 will be determined
Immunogenicity of QLF31907 | up to 2 years
  the anti-drug antibody(ADA) against QLF31907 will be determined
overall survival(OS) | up to 2 years
  the OS of QLF31907 combination therapy will be determined
maximum plasma concentration (Cmax) of QLF31907 | up to 2 years
  the maximum plasma concentration (Cmax) of QLF31907 will be determined